CLINICAL TRIAL: NCT00330460
Title: A Randomized, Double-Blind Study to Compare the Efficacy of Treatment With Denosumab Versus Alendronate Sodium in Postmenopausal Women With Low Bone Mineral Denisty
Brief Title: A Randomized, Double-Blind Study to Compare the Efficacy of Treatment With Denosumab Versus Alendronate Sodium in Postmenopausal Women With Low Bone Mineral Density.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20050141
Record Dates: First submitted 2006-04-06; First posted 2006-05-26 (Estimated); Results first posted 2010-07-19 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Osteoporosis; Osteopenia; AMG 162; Fracture - hip; Postmenopausal
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Hip Fractures | interventions — Alendronate; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Alendronate (Active Comparator): Subjects in this arm will receive active ALN and placebo denosumab
  Interventions: Drug: Alendronate
- Denosumab (Experimental): Subjects in this arm will receive active denosumab and placbo ALN
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Alendronate — ALN; 70 mg; oral; once weekly
  Arms: Alendronate
Drug: Denosumab — 60 mg; SC; every 6 months
  Arms: Denosumab

SUMMARY:
The purpose of this study is to determine whether in postmenopausal women with low bone mineral density, the mean percent change in total hip BMD in subjects receiving denosumab is not less than that observed in subjects receiving alendronate sodium by more than a pre-specified non-inferiority margin.

ELIGIBILITY:
Inclusion Criteria: - Patient is an ambulatory postmenopausal woman - Patient has BMD value that corresponds to a T-score of less than or equal to -2.0 (g/cm2) at the lumbar spine OR total hip within range specific to the study protocol. Exclusion Criteria: o Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

* Evidence of any of the following per subject report, chart review or central laboratory result:

  1. Hyper- or hypothyroidism; however, subjects on stable thyroid hormone replacement therapy may be allowed per the following criteria:

     * If TSH level is normal, subject is eligible for the study.
     * If TSH level is below normal range, subject is not eligible for the study.
     * If TSH level is elevated (> 5.5 mIU/mL to 10.0 mIU/mL), serum T4 should be measured. If serum T4 is within normal range, subject is eligible. If serum T4 is outside of normal range, subject is not eligible for the study.
     * If TSH level is above 10.0 mIU/mL, subject is not eligible.
  2. Current hyper- or hypoparathyroidism
  3. Elevated transaminases

     * Serum aspartate aminotransferase (AST; serum glutamate-oxaloacetic transaminase [SGOT]) ³ 2.0 x upper limits of normal (ULN)
     * Serum alanine aminotransferase (ALT; serum glutamate-pyruvate transaminase [SGPT]) ³ 2.0 x ULN
  4. Significantly impaired renal function as determined by serum creatinine ³ 2.0 mg/dL
  5. Current hypo- or hypercalcemia based on the central laboratory reference ranges
  6. Active gastric or duodenal ulcer; history of significant gastrointestinal bleed requiring hospitalization or transfusion, or dyspepsia or gastroesophageal reflux disease that is uncontrolled by medication
  7. Rheumatoid Arthritis, Paget's disease, Cushing's disease, hyperprolactinemia, or cirrhosis of the liver
  8. Known to have tested positive for human immunodeficiency virus, hepatitis C virus, or hepatitis B surface antigen
  9. Malignancy (except fully resected cutaneous basal cell or squamous cell carcinoma, cervical or breast ductal carcinoma in situ) within the last 5 years
  10. Any metabolic bone disease, eg, osteomalacia or osteogenesis imperfecta, which may interfere with the interpretation of the findings
  11. Malabsorption syndrome or any gastrointestinal disorders that are associated with malabsorption
* Received any solid organ or bone marrow transplant
* Vitamin D deficiency (25(OH) vitamin D level < 12 ng/mL). Vitamin D repletion will be permitted and subjects may be re-screened; see Section 7.
* Any laboratory abnormality which, in the opinion of the investigator, will prevent the subject from completing the study or interfere with the interpretation of the study results
* Contraindicated or poorly tolerant of ALN therapy; contraindications for ALN therapy include:

  1. Abnormalities of the esophagus, which delay esophageal emptying such as stricture or achalasia.
  2. Inability to stand or sit upright for at least 30 minutes.
  3. Hypersensitivity to ALN or other constituents of ALN tablets o Known sensitivity to mammalian cell derived drug products
* Known intolerance to calcium supplements
* Administration of intravenous bisphosphonate, or fluoride (except for dental treatment) or strontium ranelate
* Oral bisphosphonate treatment:

  * ³ 3 months cumulatively in the past 2 years, OR
  * ³ 1 month in the past year, OR
  * Any use during the 3-month period prior to randomization
* PTH or PTH derivatives (eg, teriparatide) within the last year
* Administration of any of the following treatments within 3 months of randomization:

  1. Any SERM (eg, raloxifene)
  2. Tibolone
  3. Anabolic steroids or testosterone
  4. Glucocorticosteroids (³ 5 mg prednisone equivalent per day for more than 10 days)
  5. Systemic (oral, transdermal, topical) hormone replacement therapy (local vaginal estrogen preparation will be allowed)
  6. Calcitonin
  7. Calcitriol or vitamin D derivatives
  8. Other bone active drugs including anti-convulsives (except benzodiazepines) and heparin
  9. Chronic systemic ketoconazole, androgens, ACTH, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, gonadotropin-releasing hormone agonists
  10. Height, weight or girth which may preclude accurate DXA measurements
* Less than 2 lumbar vertebrae (L1-L4) evaluable for DXA measurements
* Both hips not evaluable by DXA (eg, history of bilateral hip replacement or pins in both hips)
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s)
* Any physical or psychiatric disorder which, in the opinion of the investigator, will prevent the subject from completing the study or interfere with the interpretation of the study results
* Evidence of alcohol or substance-abuse within the last 12 months which the investigator believes would interfere with understanding or completing the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Brown JP, Prince RL, Deal C, Recker RR, Kiel DP, de Gregorio LH, Hadji P, Hofbauer LC, Alvaro-Gracia JM, Wang H, Austin M, Wagman RB, Newmark R, Libanati C, San Martin J, Bone HG. Comparison of the effect of denosumab and alendronate on BMD and biochemical markers of bone turnover in postmenopausal women with low bone mass: a randomized, blinded, phase 3 trial. J Bone Miner Res. 2009 Jan;24(1):153-61. doi: 10.1359/jbmr.0809010. PMID 18767928
- [Derived] Gold DT, Horne R, Coon CD, Price MA, Borenstein J, Varon SF, Satram-Hoang S, Macarios D. Development, reliability, and validity of a new Preference and Satisfaction Questionnaire. Value Health. 2011 Dec;14(8):1109-16. doi: 10.1016/j.jval.2011.06.010. Epub 2011 Oct 1. PMID 22152181
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_49_AMG_162_20050141.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 26-Apr-2006 Last Subject Enrolled: 17-Nov-2006
Period: Overall Study
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Started | 595 | 594
Completed | 553 | 561
Not Completed | 42 | 33
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 10 | 8
Not completed — Withdrawal by Subject | 18 | 17
Not completed — Death | 1 | 1
Not completed — Ineligibility determined | 1 | 3
Not completed — Lost to Follow-up | 8 | 3
Not completed — Noncompliance | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M | Total
Number analyzed (Participants) | 595 | 594 | 1189
Age Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (8.3) | 64.1 (8.6) | 64.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 595 | 594 | 1189
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 502 | 502 | 1004
  Black or African American | 9 | 7 | 16
  Hispanic or Latino | 69 | 66 | 135
  Asian | 8 | 6 | 14
  Japanese | 4 | 3 | 7
  American Indian or Alaska Native | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Population: Randomized subjects who have a nonmissing baseline and at least 1 nonmissing postbaseline evaluation at or prior to month 12. LOCF used as imputation method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 572 | 579
Percent Change from Baseline | 2.6 [2.4 to 2.8] | 3.5 [3.3 to 3.7]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -1.22%; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1, 95% CI [0.7 to 1.2]

2. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 571 | 579
Percent Change from Baseline | 4.2 [3.9 to 4.5] | 5.3 [5.0 to 5.6]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -2.29%; p < 0.0001, ANCOVA — The reported p-value was the one-sided adjusted p-valued based on multiplicity adjustment of the secondary efficacy endpoints; Mean Difference (Final Values) = 1.1, 95% CI [0.7 to 1.4]

3. Secondary Outcome: Trochanter Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 572 | 579
Percent Change from Baseline | 3.4 [3.1 to 3.7] | 4.5 [4.1 to 4.8]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -1.65%; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1, 95% CI [0.6 to 1.4]

4. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 572 | 579
Percent Change from Baseline | 1.8 [1.5 to 2.1] | 2.4 [2.2 to 2.7]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -1.04%; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI [0.3 to 1]

5. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 569 | 573
Percent Change from Baseline | 0.6 [0.3 to 0.8] | 1.1 [0.9 to 1.4]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI [0.3 to 0.9]

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 37/586 | 34/593
Other Adverse Events (participants affected / at risk) | 261/586 | 270/593
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alendronate 70 mg QW (N=586) | Denosumab 60 mg Q6M (N=593)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Ventricular asystole (Cardiac disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 3
Ear infection (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Pelvic peritoneal adhesions (Reproductive system and breast disorders) | 1 | 0
Urogenital prolapse (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Activities of daily living impaired (Social circumstances) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alendronate 70 mg QW (N=586) | Denosumab 60 mg Q6M (N=593)
Constipation (Gastrointestinal disorders) | 31 | 36
Diarrhoea (Gastrointestinal disorders) | 20 | 30
Dyspepsia (Gastrointestinal disorders) | 29 | 34
Influenza (Infections and infestations) | 42 | 41
Nasopharyngitis (Infections and infestations) | 43 | 45
Upper respiratory tract infection (Infections and infestations) | 25 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 56 | 75
Back pain (Musculoskeletal and connective tissue disorders) | 56 | 42
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 31
Headache (Nervous system disorders) | 32 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.